CLINICAL TRIAL: NCT06638294
Title: A Translational Observational Biorepository and Management Study in Patients With Breast Cancer Leptomeningeal Metastasis: The BioLept Study
Brief Title: Study in Patients With Breast Cancer Leptomeningeal Metastasis
Acronym: BioLept
Status: Recruiting | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Avon Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: J2323; IRB00371039 (Other: Johns Hopkins IRB)
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Leptomeningeal Metastasis of Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cerebrospinal fluid (CSF) collections and blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with breast cancer leptomeningeal disease (LMD): Participation involves allowing access to participant medical records including the genetic information of the tumor, undergoing standard-of-care work up as indicated (this may include MRI of brain or spine, spinal tap, etc.), providing a cerebrospinal (CSF) sample (less than 2 tablespoons), blood sample (about 4 tablespoons) at baseline and possibly again after month, and answering online questionnaires monthly.
  Johns Hopkins Molecular Tumor Board will review clinical and genetic information and provide treatment recommendations. CSF and blood will be collected at baseline no matter what treatment is recommended. If possible, collect CSF and blood again after one month. Additional blood and CSF sampling may also be obtained if/when therapy changes.
  The oncologist will ultimately decide if participant will proceed with the recommend treatment or not. Health information and questionnaires are obtained to assess how participants are doing on therapy.

SUMMARY:
Traditional clinical trials in patients with breast cancer leptomeningeal disease (LMD) are challenging as patients often have a rapidly progressive course and prognosis is poor, making meeting standard eligibility difficult. Furthermore, there is limited information about the biology of LMD. The investigators thus propose a study that is as inclusive as possible, which will allow the investigators to collect biospecimens and clinical outcomes to learn more about LMD biology, but still potentially provide benefit for patients, by providing patients rapid diagnostics and multi-disciplinary treatment recommendations.

DETAILED DESCRIPTION:
This is a prospective translational observational study for patients with breast cancer leptomeningeal disease (LMD). LMD is notoriously difficult to treat, and prognosis is generally very poor, with most patients typically succumbing to the disease within a few months of its diagnosis. Conducting clinical trials is challenging for these reasons, and there are limited data regarding biological processes of LMD. The overarching goal of this study is to be as inclusive as possible to optimize and learn from patients with LMD. The investigators propose a prospective observational study to establish (1) a translational collection protocol to comprehensively collect tissue, blood, and CNS samples, and (2) a therapeutic management program utilizing the Johns Hopkins Molecular Tumor Board, to provide multi-disciplinary treatment recommendations in a timely manner, and (3) collect outcome data that can be correlated with biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 or older
* History of breast cancer (any subtype)
* Suspected breast cancer-related leptomeningeal metastasis (i.e., by clinical signs or symptoms (i.e., peri-oral dysesthesia, unexplained new neurological symptoms in the absence of brain metastasis), radiographic, or by cerebrospinal fluid analysis), whereby patient will be treated along an leptomeningeal disease paradigm.
* Previous central nervous system metastasis (including leptomeningeal disease or brain metastasis) is eligible.
* Eastern Cooperative Oncology Group (ECOG) score of ≤3 or Karnofsky performance status ≥60.

Exclusion Criteria:

* Suspected central nervous system recurrence of hematologic malignancy, lymphoma or other solid tumor
* Not eligible for treatment of leptomeningeal disease.

Min Age: 18 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a prospective translational observational study for patients with breast cancer leptomeningeal disease (LMD).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who achieve goal time to treatment recommendation | 2 years
  Rapid molecular tumor board (MTB) evaluation. The investigators will measure the percentage of patients who achieve the following the goal time to treatment recommendation. The investigators goal time to treatment recommendation will be ≤7 days from enrollment, and the investigators goal time to treatment initiation ≤14 days from enrollment.
  There is no set goal in terms of percentage of patients achieving set timeframes as there will be a significant variability. The investigators hope to continuously refine this process to meet these ideal timeframes. The investigators will report the investigators' ability to achieve these timeframes in order to evaluate the feasibility of rapid molecular tumor board (MTB) evaluation and time to treatment in patients with breast cancer leptomeningeal disease (LMD)..

SECONDARY OUTCOMES:
Correlation of patient reported outcomes and biomarkers | 2 years
  The investigators will assess patient reported outcomes (PROs) using the Patient-Reported Outcomes Measurement Information System Global-10 (PROMIS Global-10) and select questions from the Functional Assessment of Cancer Therapy - Central nervous System (FACT-CNS) and Functional Assessment of Cancer Therapy-Brain (FACT-Br) questionnaire. The investigators will describe development of central nervous systems and clinical deterioration, and correlate with patient reported outcomes and biomarkers including Germline testing and Tumor Next Generation Sequencing.
Correlation of molecular features of cerebrospinal fluid and cerebrospinal fluid biomarkers | 2 years
  Molecular features of cerebrospinal fluid (CSF) including circulating tumor cell (CTCs) and cell-free tumor DNA (ctDNA). Cerebrospinal fluid biomarkers will be described and correlated with standard CSF assessments including cytology and cell count, radiographic assessments, and clinical outcomes, and correlate these with standard CSF and radiographic assessments, and patient outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Cesar Santa-Maria, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (2):
- United States (2):
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland